CLINICAL TRIAL: NCT04919291
Title: Contralateral Comparison of Togoguided LASIK and Wavefront-optimized LASIK
Brief Title: Direct Comparison of TG and WFO LASIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Nobel Eye Clinic (Other)
Responsible Party: Principal Investigator, Chao-Kai Chang, Dean, Nobel Eye Institute, Taipei Nobel Eye Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2021-03-23; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Keratomileusis, Laser In Situ; Contrast Sensitivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topoguided LASIK (Active Comparator): Topoguided ablation profile on dominant eye
  Interventions: Device: Topoguided LASIK
- Wavefront optimized LASIK (Active Comparator): Wavefront optimized ablation profile on non-dominant eye
  Interventions: Device: Wavefront optimized LASIK

INTERVENTIONS:
Device: Topoguided LASIK — Topoguided ablation profile on dominant eye
  Arms: Topoguided LASIK
Device: Wavefront optimized LASIK — Wavefront optimized ablation profile on non-dominant eye
  Arms: Wavefront optimized LASIK

SUMMARY:
To compare the efficacy to different profiles, direct head-to-head studies had been conducted. In one previous review study revealed that TG LASIK provided patient with better uncorrected visual acuity (UCVA) than WFO LASIK and WFG LASIK. In recent previous contralateral eye studies also showed that TG LASIK induced less postoperative higher-order aberration than WFO LASIK. However, these studies included only low-to-moderate myopia patients, for patients with high myopia (spherical equivalent > 6D), the effect of TG LASIK comparing with WFO LASIK had not been reported before.

The aim of our study is to analyze and compare the visual performance of TG LASIK and WFO LASIK in high myopia and low-to-moderate myopia patients, , particularly UCVA, corrected distance visual acuity (CDVA), contrast sensitivity (CS), and wavefront aberration.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 50 years old
* CDVA of both eyes could reach 0.1 logarithm of the minimum angle of resolution (logMAR)
* stable refractive errors of myopia and astigmatism

Exclusion Criteria:

* cataract
* corneal opacities or irregularities
* dry eye (Schirmer's test I ≤ 5mm)
* amblyopia
* coexisting ocular pathologies
* glaucoma
* non-dilating pupil
* history of intraocular surgery, laser therapy, or retinopathy
* optic nerve or macular diseases
* estimated postoperative cornea residual stromal thickness less than 250 μm
* pregnancy or under lactation
* uncontrolled diabetic mellitus or systemic immune disease
* refusal or unable to maintain follow-up

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 3 months after surgery
  uncorrected visual acuity and corrected distance visual acuity
Corneal wavefront analysis | 3-months postoperative visit
  horizontal coma aberration (Z 3,1), spherical aberration (Z 4,0), and trefoil aberration
Contrast sensitivity | 3-months postoperative visit
  4 spatial frequencies: 3, 6, 12, and 18 cycles per degree (cpd).
Quality of vision questionnaire | 3-months postoperative visit
  A 11-item questionnaire, item scores range from 0 to 10 and higher item scores in questionnaire indicated more difficulty in achieving specific visual tasks

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Nobel Eye Clinic, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sutton G, Lawless M, Hodge C. Laser in situ keratomileusis in 2012: a review. Clin Exp Optom. 2014 Jan;97(1):18-29. doi: 10.1111/cxo.12075. Epub 2013 Jun 21. PMID 23786377
- [Background] Moreno-Barriuso E, Lloves JM, Marcos S, Navarro R, Llorente L, Barbero S. Ocular aberrations before and after myopic corneal refractive surgery: LASIK-induced changes measured with laser ray tracing. Invest Ophthalmol Vis Sci. 2001 May;42(6):1396-403. PMID 11328757
- [Background] Schallhorn SC, Farjo AA, Huang D, Boxer Wachler BS, Trattler WB, Tanzer DJ, Majmudar PA, Sugar A; American Academy of Ophthalmology. Wavefront-guided LASIK for the correction of primary myopia and astigmatism a report by the American Academy of Ophthalmology. Ophthalmology. 2008 Jul;115(7):1249-61. doi: 10.1016/j.ophtha.2008.04.010. PMID 18598819
- [Background] Stonecipher K, Parrish J, Stonecipher M. Comparing wavefront-optimized, wavefront-guided and topography-guided laser vision correction: clinical outcomes using an objective decision tree. Curr Opin Ophthalmol. 2018 Jul;29(4):277-285. doi: 10.1097/ICU.0000000000000495. PMID 29787391
- [Background] Kim J, Choi SH, Lim DH, Yang CM, Yoon GJ, Chung TY. Topography-guided versus wavefront-optimized laser in situ keratomileusis for myopia: Surgical outcomes. J Cataract Refract Surg. 2019 Jul;45(7):959-965. doi: 10.1016/j.jcrs.2019.01.031. Epub 2019 Jun 10. PMID 31196580
- [Background] Kim J, Choi SH, Lim DH, Yoon GJ, Chung TY. Comparison of outcomes after topography-modified refraction versus wavefront-optimized versus manifest topography-guided LASIK. BMC Ophthalmol. 2020 May 14;20(1):192. doi: 10.1186/s12886-020-01459-0. PMID 32410588
- [Background] Ozulken K, Yuksel E, Tekin K, Kiziltoprak H, Aydogan S. Comparison of Wavefront-Optimized Ablation and Topography-Guided Contoura Ablation With LYRA Protocol in LASIK. J Refract Surg. 2019 Apr 1;35(4):222-229. doi: 10.3928/1081597X-20190304-02. PMID 30984979